CLINICAL TRIAL: NCT03352440
Title: The Use of Different Devices Through Virtual Reality in People With Cerebral Palsy
Brief Title: Different Virtual Reality Devices in People With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Carlos Bandeira de Mello Monteiro, Associate Professor, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 32476414.5.0000.0082
Record Dates: First submitted 2017-11-17; First posted 2017-11-24 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Virtual Reality Exposure Therapy; Learning; Motor Activity; Motor Skills
MeSH Terms: conditions — Cerebral Palsy; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cerebral Palsy - Kinect (Experimental): Group with Cerebral Palsy that will perform the task on Kinect
  Interventions: Device: Cerebral Palsy - Kinect
- Cerebral Palsy - Touchscreen (Experimental): Group with Cerebral Palsy that will perform the task on Touchscreen
  Interventions: Device: Cerebral Palsy - Touchscreen
- Control Group - Kinect (Active Comparator): Group with typical development that will perform the task on Kinect
  Interventions: Device: Control Group - Kinect
- Control Group - Touchscreen (Active Comparator): Group with typical development that will perform the task on Touchscreen
  Interventions: Device: Control Group - Touchscreen

INTERVENTIONS:
Device: Cerebral Palsy - Kinect — Group with Cerebral Palsy that will perform the task on Kinect
  Arms: Cerebral Palsy - Kinect
Device: Cerebral Palsy - Touchscreen — Group with Cerebral Palsy that will perform the task on Touchscreen
  Arms: Cerebral Palsy - Touchscreen
Device: Control Group - Kinect — Group with typical development that will perform the task on Kinect
  Arms: Control Group - Kinect
Device: Control Group - Touchscreen — Group with typical development that will perform the task on Touchscreen
  Arms: Control Group - Touchscreen

SUMMARY:
A computer program was developed with the same task, but with two possibilities of user interaction: a) interface with contact: in which the individual touches the computer screen to finish the task and b) interface without contact: in which the individual perform a hand movement in front of the Kinect. Were evaluated 29 individuals with CP who constituted the experimental group and 28 individuals without deficiency who composed the control group with matching age and sex.

DETAILED DESCRIPTION:
A total of 57 individuals were included in this study, 29 individuals with CP who constituted the experimental group and 28 individuals without deficiency, aged between 6 and 15 years, with understanding of the task to be performed. Of these, 14 formed the experimental group 1 that performed the task on Kinect (CP-Group1) and 15 individuals formed the control group 1 (TD-Group1), 15 formed the experimental group 2 (CP-Group2) and 13 individuals formed the control group 2 (TD-Group2), all control groups matched for age and sex with the experimental group 1 and 2, all without any disability.

All individuals with CP who were evaluated manage to stay well seated to function in the upper limbs and have independent walking even necessary aid walker or crutches.

Material and Apparatus Software specialists developed a package of games, named Team Bridge Games, and for this study, was used the Check Limit Game. This game allows the use of a Kinect sensor for motion capture (without contact interface), as well as a touch screen (with contact interface). The virtual reality tool used was developed by the Information Systems Laboratory of EACH / USP which features on the computer a task in which several balls are on the screen and must be touched to change color. The goal is to change the maximum of balls color in 15 seconds. The touch is performed through the touch screen corresponding to the physical environment with tap or by means of touchless environment using a virtual interface offered by Kinect system. Data regarding performance will be analyzed considering the number of hit balls.

Procedure and Design To perform the task virtual research participants will be positioned at the computer so that they are adjusted in height (this will depend on the physical composition of each participant) and away from the computer screen, approximately 1.5m., and also the interface used thus enabling the beginning of the task.

It were previously explained to the participant as it should do it with the Kinect, which through actual movement the individual has the ability to perform a task, using an avatar, each with their specific implementation, with one of the upper limbs and fingers of one hand respectively; should be aware of the start of the task as the verbal command of the researcher, for each phase of the task to be performed has duration of 7 minutes and 30 seconds, 1 minute and 15 seconds respectively, with five-minute interval, consisting of the acquisition phase ( the activity will be repeated 30 times / attempts), retention (will repeat the activity 5 times / attempts) and transfer (activity will be repeated 5 times / attempts) respectively.

Considering an estimated running time of approximately 30 minutes in just one meeting. Both the experimental group and the control group performed two tasks: real and virtual environment, where the control and experimental group-1 performed the following sequence: Acquisition = Kinect, Retention = Kinect and Transfer = Touchscreen; the experimental control group-2 and performed the following sequence: Acquisition = Touchscreen, Retention = Touchscreen and Transfer = Kinect.

ELIGIBILITY:
Inclusion Criteria:

* individuals with a diagnosis PC (for the experimental group);
* diparesis and spastic hemiparesis;
* with gross motor function classification as levels I, II and III according to the Gross Motor Function Classification System (GMFCS).

Exclusion Criteria:

* individuals who have undergone surgery or performing chemical neuromuscular blockade for less than 6 months in the upper limbs;
* associated diseases;
* changes in cognitive functions that preclude cooperation and understanding in the proposed activities.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Improvement of performance on Touchscreen interface provided by the Kinect system. | one day
  The number of bubbles reached with the attempts will show the improvement of performance.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos BM Monteiro, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Escola de Artes,Ciencias e Humanidades da Universidade d Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Leal AF, da Silva TD, Lopes PB, Bahadori S, de Araujo LV, da Costa MVB, de Moraes IAP, Marques RH, Crocetta TB, de Abreu LC, Monteiro CBM. The use of a task through virtual reality in cerebral palsy using two different interaction devices (concrete and abstract) - a cross-sectional randomized study. J Neuroeng Rehabil. 2020 Apr 29;17(1):59. doi: 10.1186/s12984-020-00689-z. PMID 32349752